CLINICAL TRIAL: NCT02473549
Title: Towards More Successful Clinical Trials: Using a Patient-tailored Approach in Brain Stimulation to Improve Recovery of Movements After Stroke
Brief Title: Improving Motor Stroke Recovery Using Patient-tailored Non-invasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 143-2015
Record Dates: First submitted 2015-05-25; First posted 2015-06-16 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Stroke
Keywords: motor; rehabilitation; transcranial direct current stimulation
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brain Stimulation (Experimental): Patients will receive, Sham TDCS, Anodal TDCS, Cathodal TDCS, and Magnetic Resonance Imaging (MRI).
  Interventions: Device: Sham TDCS; Device: Anodal TDCS; Device: Cathodal TDCS; Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Sham TDCS — Placebo stimulation is applied to the unaffected motor cortex while participants perform rehabilitation exercises for the upper extremity
Device: Anodal TDCS — Excitatory stimulation is applied to the unaffected motor cortex while participants perform rehabilitation exercises for the upper extremity
Device: Cathodal TDCS — Inhibitory stimulation is applied to the unaffected motor cortex while participants perform rehabilitation exercises for the upper extremity
Device: Magnetic Resonance Imaging (MRI) — Participants will receive a MRI of their brain to allow the research investigators to determine how the stroke has affected regions of the brain processing movements.

SUMMARY:
Many individuals are often left with problems moving their arm and hand, months to even years after a stroke. Recent progress in research suggests the application of non-invasive brain stimulation, such as transcranial direct current stimulation (TDCS), in conjunction with rehabilitation exercises can further improve a person's ability to move after stroke. However, the problem is that this doesn't work for everyone, and researchers do not know why. One reason may be that TDCS is currently applied using a one-size-fits-all approach. Researchers apply the same type of TDCS to everyone, assuming the stroke affects everyone in the same way. But, researchers know this is not the case. For example, each person will likely have different amounts of damage to brain regions that control movements. A better understanding of how the stroke uniquely affects a person's brain will help us to know which is the correct type of TDCS to apply for that person. Therefore, the objective of this research is to determine whether the amount of damage to brain regions that control movements can predict which type of TDCS will be more effective to help a person improve their ability to move. Participants will undergo 1 session of magnetic resonance imaging, and three sessions of TDCS.

ELIGIBILITY:
Inclusion Criteria:

* unilateral first time stroke in middle cerebral artery territory
* greater 3 months post-stroke
* able to raise arm onto a table from a seated position

Exclusion Criteria:

* severe cognitive or comprehension deficits that may compromise informed consent or understanding of instructions
* severe apraxia and neglect
* neurodegenerative or psychiatric disease
* contraindications to MRI and TDCS (e.g. metal in head, pacemaker, claustrophobia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in movement time (seconds) for reaching after 1 session of TDCS | 1 day
Change in accuracy of reaching (root mean square error) after 1 session of TDCS | 1 day
Change in efficiency of reaching (number of velocity peaks) after 1 session of TDCS | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chen, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada